CLINICAL TRIAL: NCT06310681
Title: A Co-adapted Community-based Participatory Group Programme for Parents/Carers of Children With Complex Neurodisability (ENCOMPASS): A Pilot and Feasibility Study
Brief Title: Pilot Testing of a Co-adapted Group Programme for Parents/Carers of Children With Complex Neurodisability
Acronym: ENCOMPASS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ETH2223-2528
Record Dates: First submitted 2024-02-27; First posted 2024-03-15 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Complex Neurodevelopmental Disorder; Cerebral Palsy
Keywords: Community-based programme; cerebral palsy; caregiver; parent; peer support; feasibility; acceptability; children; complex neurodisability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Encompass" group programme (Experimental)
  Interventions: Behavioral: "Encompass" group programme

INTERVENTIONS:
Behavioral: "Encompass" group programme — * Groups will take place over ten modules
  * They will take place in-person at a local community venue
  * The groups will be two hours long, with a break for refreshments in the middle. They will take place every fortnight in term-time only over approximately 6 months.
  * The groups predominantly follow a participatory learning approach and although the facilitators have manuals, the activities tend to include some imparting of information, key points for discussion, examples from other settings and activities for the group to practice.
  * They are run by two facilitators - one parent with lived experience and one healthcare professional

SUMMARY:
The goal of this pilot feasibility study is to test a co-adapted community-based group programme ("Encompass") with parents/carers of children with complex neurodisability under 5 years of age in East London in the UK.

The main questions it aims to answer are:

* Is it feasible and acceptable to carry out this newly co-adapted programme with two groups of parents/carers of children with complex neurodisability under the age of 5?
* Is it feasible to carry out an evaluation of the above programme, which could then inform a protocol for larger scale evaluation?

The main activities for the parent/carer participants will include:

* Attending ten "Encompass" parent/carer groups
* Filling in questionnaires at the start and end of the groups
* Attending an interview with the researcher to discuss their experiences

The groups will be facilitated by a healthcare professional and a parent with lived experience. They will also be interviewed about their experiences after the groups have been completed.

DETAILED DESCRIPTION:
Background

Parents/carers of children with complex neurodisability continue to lack appropriate family-centred care. "Encompass" is a community-based group programme that was co-adapted from "Baby Ubuntu" in Uganda. It is an example of a 'decolonised healthcare innovation' as it is a low-cost solution from a low-income country for use in a resource-constrained UK National Health Service (NHS).

Methods and analysis

The investigators will conduct a mixed methods pilot feasibility study to determine the feasibility and acceptability of delivering and evaluating "Encompass" with parents/carers of children under 5 years with complex neurodisability in the UK. The investigators aim to recruit 20 parents/carers of children from two NHS trusts in England serving urban areas where there is high social deprivation and ethnic diversity. Recruited parents/carers will attend the 10-modular, participatory group programme over a 6-month period. Groups will be facilitated by a trained allied health professional and an 'expert parent' with lived experience. The primary outcomes of interest are the feasibility of delivering and evaluating the programme (recruitment, retention rates, acceptability as perceived by the parents/carers, facilitators and wider key stakeholders), intervention fidelity and participant adherence. Results will be collectively assessed against traffic light criteria. Pre-, post- and follow-up data collection questionnaires will include the Family Empowerment Scale (FES), the Power Ladder Question, the Parent Patient Activation Measure (P-PAM), Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS), EuroQoL-5D-5-level (EQ-5D-5L) and parent/carer greatest needs and goals questionnaire. Post-intervention semi-structured interviews will be conducted with parents/carers, facilitators and key stakeholders within the NHS.

Discussion

Providing family-centred support through a community-based participatory group programme is a potentially affordable and sustainable way for the NHS to improve a range of outcomes for parents/carers of children with complex neurodisability including knowledge, skills and confidence, wellbeing and quality of life. The programme also provides opportunities for peer support and aims to empower parents/carers in navigating community health systems.

ELIGIBILITY:
Parents and carers:

Inclusion Criteria:

* Care for a child (<5 years) with a complex neurodisability*
* Have received a diagnosis for their child, which has been disclosed to them, even this is a diagnosis such as SWAN (Syndrome Without A Name)
* Reside in the boroughs of Newham or Tower Hamlets, East London
* ≥18 years of age.

Exclusion Criteria:

* Have a child with a developmental disability where there are no functional physical impairments as part of their complex needs. For example, children diagnosed with Autism Spectrum Disorder, Attention Deficit Hyperactivity Disorder, intellectual impairments will be excluded unless they have a functional physical impairment with a neurological cause too.
* Have a child with a progressive neurological condition such as Duchenne's Muscular Dystrophy.
* Have a child with a structural physical impairment not caused by a neurological event or neurological difficulties. For example, children born with a limb difference or a child with hearing loss.
* Do not have capacity to consent
* Do not meet the inclusion criteria as specified above
* There are no exclusions based on language, as interpreting/translating services will be offered.

Parent Facilitator:

Inclusion Criteria:

* Parents/carer of children with complex neurodisability who are identified through other services as potentially being able to facilitate a group as an 'expert parent'
* Prior experience in training or using participatory approaches - not essential

Exclusion Criteria:

* Inability to read and speak English
* Inability to commit to a 6-month period of work to the best of their knowledge

Healthcare Professional Facilitator:

Inclusion Criteria:

* Therapists or healthcare professionals who work with children with disabilities and who are open to learning with families about their children.
* Need to be registered with the Health and Care Professionals Council and should ideally have > 5 years post-graduate experience working with a paediatric population
* Confident in working with children with complex neurodisability, such as cerebral palsy

Exclusion Criteria:

* Inability to read and speak English
* Inability to commit to a 6-month period of work to the best of their knowledge

Key Stakeholders:

Inclusion Criteria:

* Staff from the NHS that are either involved in the delivery or commissioning of community child health care services in Newham or Tower Hamlets.
* Examples include clinical managers, service leads or commissioners.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Group Attendance | End of each group, 6 months
  Green light - More than 80% of parents/carers attend the group for 6+ sessions Amber light - 30-79% of parents/carers attend the group for 6+ sessions Red light - Fewer than 30% attend the group for 6+ sessions
  Feasibility, acceptability, and process outcome measures will be used. Quantitative data will be collected to assess the Traffic Light criteria. The green light signifies that criteria for progression has been met and a larger evaluation could proceed, the amber light suggests certain amendments need to be made and the red light indicates that the criteria for progression have not been met and researchers should not continue to a trial.
Recruitment - percentage of eligible participants who consent to take part | Before the groups commence, 3 months
  Green light - 35% who are eligible consent to participate Amber light - 15-34% who are eligible consent to participate Red light - Less than 15% who are eligible consent to participate
Follow-up response rate-self-complete outcomes questionnaire(s) | Through the groups and 3 months post-groups, approximately 9 months
  Green light - 70% or greater response to follow up Amber light - 50-69% response to follow up Red light - Less than 50% response to follow up
Fidelity - delivery on items described in the Fidelity Checklist | End of each group, 6 months
  Green light - 70% or greater score on the checklist Amber light - 50-69% score on the checklist Red light - Less than 50% score on the checklist

SECONDARY OUTCOMES:
Family Empowerment Scale (FES) | First and final groups, 6 months
  The Family Empowerment Scale (FES) is a validated 24-item instrument that measures parents' sense of empowerment across three areas; family, service use and community. It has been used in the ENVISAGE (ENabling VISions And Growing Expectations) parent workshops and aligns with the goals of the 'Encompass' groups which are to empower families to understand their child's diagnosis and how to navigate health systems. A limitation of this tool is that it has mostly been used with a white, US population.
Power Ladder Question (PLQ) | First and final groups, 6 months
  The Power Ladder Question (PLQ) assesses participants' perceived sense of power and influence over their life. The survey asks "Please imagine a nine-step ladder, where on the bottom, the first step, stand people who are completely without rights, and on the highest step, the ninth, stand those who have a lot of power. On which step are you?". It has been used with diverse groups and allows the participant to choose the domains of power that they value, and interpret the question openly.
Parent Patient Activation Measure (P-PAM) | First and final groups, 6 months
  Parent patient activation relates to the knowledge, skills, confidence and persistence to manage a child's health care, particularly those with developmental disorders or disabilities. The Parent-Patient Activation Measure (P-PAM) is a validated 13-item tool that measures two factors; 'confidence and knowledge' and 'action and perseverance' . It has been used in a variety of diverse settings, including low income, non-English speaking parents.
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | First and final groups, 6 months
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) has been widely used to assess wellbeing across a diverse range of public health interventions, populations, and settings. The 14-item scale WEMWBS will be used with 5 response categories that are summed up to provide a single score.
Parent/carer Quality of Life - EuroQoL-5D-5-level (EQ-5D-5L) | First and final groups, 6 months
  The EuroQoL five-dimension questionnaire is a validated and widely used tool that measures generic quality of life. It has one question for each of the five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with five response options
Parent/carer Needs and Goals | First group, 1 month
  A questionnaire has been adapted from previous evaluations of Ubuntu interventions. It has two questions and asks parents/carers what their three biggest issues are that they face in everyday life, and what their two main goals are for attending the group.
Childhood Cost Calculator (C3) | End of study, 9 months
  A costing tool for education and early childhood development.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Barts Health NHS Trust, Children's Occupational Therapy, Mile End Hospital, London
  - East London NHS Foundation Trust, Specialist Children's and Young People's Services, London

REFERENCES:
- [Derived] Prest K, Harden A, Barnicot K, Heys M. A coadapted community-based participatory group programme for parents/carers of children with complex neurodisability (Encompass-2): a pilot and feasibility study protocol. Pilot Feasibility Stud. 2025 May 3;11(1):59. doi: 10.1186/s40814-025-01619-3. PMID 40319319
- See also: Encompass Study website — https://www.encompassresearch.org/